CLINICAL TRIAL: NCT04679896
Title: A Prospective, Randomized, Single-center Study to Assess the Performance of MagnetOs Putty Compared to Local Autograft in Patients Undergoing up to Three-level Instrumented Posterolateral Lumbar Fusion (PLF).
Brief Title: Post Marketing Study of MagnetOs Putty Compared to Local Autograft in Patients Undergoing Posterolateral Lumbar Fusion
Acronym: PARTNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Collaborators: Orthopaedic Institute of Western Kentucky (Unknown); Simplified Clinical Data Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAG-920-059
Record Dates: First submitted 2020-12-18; First posted 2020-12-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Degenerative Disc Disease; Spine Fusion
Keywords: Degenerative Disc Disease; Spine Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Intra-patient control. Each patient serves as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MagnetOs Putty (Experimental): MagnetOs Putty use in instrumented posterolateral fusion, 7cc-10cc mixed with autograft bone in a 1:1 ratio per spine level at the randomized assigned side.
  Interventions: Device: MagnetOs Putty
- Local autograft (Other)
  Interventions: Device: MagnetOs Putty

INTERVENTIONS:
Device: MagnetOs Putty — Procedure: Instrumented posterolateral spine fusion

SUMMARY:
This is a phase IV post-marketing study for MagnetOs Putty. MagnetOs Putty is a synthetic bone graft extender product that is routinely used by surgeons as a treatment for patients with leg pain and/or back pain and undergoing spinal fusion surgery.

In this study, MagnetOs Putty will be used according to the latest U.S. Instructions For Use, specifically as a bone graft extender mixed with autograft in a 1:1 vol.% in the posterolateral spine.

DETAILED DESCRIPTION:
In this study, following a screening period of a maximum of 30 days, 30 patients will undergo up to a three-level instrumented posterolateral fusion (PLF) procedure. Prior to surgery, each patient will be randomized to receive MagnetOs Putty on the assigned side of the spine and local autograft bone on the other at the diseased levels. They will be followed up at discharge, Week 2, Week 6, Month 3, Month 6, and Month 12. An interim analysis will be performed once 15 patients have completed their Month 6 visit and have measurements for the endpoints available to measure effectiveness. The primary endpoint will be analyzed at Month 12.

In this study, MagnetOs Putty will be applied according to the latest Instructions for Use approved in the United States. Specifically, MagnetOs Putty will be used as a bone graft extender mixed with autograft in a 1:1 vol.% in patients with with leg pain and/or back pain requiring up to three-level instrumented posterolateral lumbar fusion procedure. The fusion procedure (PLF) will be left to the surgeon's discretion.

Radiographs will be obtained at Screening, Day 0, Week 6, Month 3. CT scans will only be obtained at Month 6 and Month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to read/be read, understand, and provide written informed consent and has signed the Investigational Review Board (IRB) approved informed consent.
2. Male or female patient ≥ 18 years old.
3. Patients with leg pain and/or back pain requiring up to three-level instrumented posterolateral lumbar fusion (L2 - S1).
4. Failed conservative treatment (physical therapy, bed rest, medications, spinal injections, manipulations, or transcutaneous electrical nerve stimulation) for a minimum period of 3 months prior to study enrollment.

Exclusion Criteria:

1. Requires > three-level fusion or expected to need secondary intervention within one year following surgery.
2. To treat conditions in which general bone grafting is not advisable.
3. In conditions where the surgical site may be subjected to excessive impact or stresses, including those beyond the load strength of fixation hardware (e.g. defect site stabilization is not possible).
4. In case of significant vascular impairment proximal to the graft site.
5. In case of severe metabolic or systemic bone disorders (e.g., osteogenesis imperfecta or Paget's Disease) that affect bone or wound healing.
6. In case of acute and chronic infections in the operated area (soft tissue infections; inflammation, bacterial bone diseases; osteomyelitis).
7. When intraoperative soft tissue coverage is not planned or possible.
8. Undergoing any procedure that allows MagnetOs to come in direct contact with the articular space.
9. Receiving treatment with medication interfering with calcium metabolism.
10. Women who are or intend to become pregnant within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Radiographic Fusion by CT Scan | Month 12
  The rate of posterolateral lumbar/thoracolumbar fusion assessed by CT-scan at Month 12. Radiographic as determined by evidence of bridging trabeculae or continuous bony connection between the superior and inferior transverse processes.

SECONDARY OUTCOMES:
Radiographic Fusion by Plain Radiographs | Week 2, Week 6, Month 3
  The rate of posterolateral lumbar fusion assessed by plain radiographs
Posterolateral lumbar fusion assessed by CT-scan | Month 6
  The rate of posterolateral lumbar fusion assessed by CT-scan at Month 6. Radiographic as determined by evidence of bridging trabeculae or continuous bony connection between the superior and inferior transverse processes
Interbody lumbar fusion assessed by plain radiographs | Week 2, Week 6, Month 3, Month 6, Month 12
  The rate of interbody lumbar fusion assessed by plain radiographs at Week 2, Week 6, Month 3, Month 6, and Month 12. Radiographic as determined by evidence of bridging trabeculae or continuous bony connection between the superior and inferior vertebral bodies
Functional Outcome by Oswestry Disability Index | Week 2, Week 6, Month 3, 6, and 12
  Change in functional score using Oswestry Disability Index questionnaire. Patient-completed survey provides subjective percentage score for level of function (disability) in activities of daily living. Score rage 0-100 percent. The lower the percentages indicate higher functionality; 0-20% minimal disability, 80-100% significant disability.
General, back and Leg Pain by Visual Analog Pain Scale | Week 2, Week 6, Month 3, 6, and 12
  Change in general, back and leg pain using Visual Analog Pain Scale score. The patient completed questionnaire is a unidimensional measure of pain intensity using a continuous scale comprised of a horizontal line 10 centimeters (100 mm) in length. The line is anchored by "no pain" (score of 0) and "worst imaginable pain". A higher score indicates greater pain intensity.
Neurologic Status by Physical Exam | Week 2, Week 6, Month 3, 6, and 12
  Change in neurologic status by examination to document stable, improved, or deficits in condition. Stable or improved findings for the lower extremities, specifically in reflexes, muscle strength, sensory, and straight leg raise.
Success Rate | Week 2, Week 6, Month 3, 6, and 12
  Number of patients with secondary surgical interventions (SSI's) such as revisions, re-operations, removals, supplemental fixations, or any other procedure that adjusts or removes part of the original implant configuration with or without replacement of the components within 12 months of surgery

OTHER OUTCOMES:
Safety Endpoint - number of patients with Adverse Events | 12 Months
  The number of patients with Adverse Events from Screening up to Month 12 after surgery
Safety Endpoint - number of patients with Serious Adverse Events | 12 Months
  The number of patients with Serious Adverse Events from Screening up to Month 12 after surgery
Safety Endpoint - number of patients with Adverse Device Effects | 12 Months
  The number of patients with Adverse Device Effects from Screening up to Month 12 after surgery
Safety Endpoint - number of patients with Device Related Complications | 12 Months
  The number of patients with any complications considered to device related with 12 months after surgery
Health Economic - Duration of Surgery | 12 Months
  Duration of surgery in minutes
Health Economic - Duration of Hospitalization | 12 Months
  Duration of hospital stay in days
Health Economic - Return to Work | 12 Months
  Time to return to work in days
Health Economic - Quality of Life | Week 6, Month 3, 6, and 12
  Change in Quality of Life measurement using EuroQol 5D/5L scoring

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Longlade, MD, Study Director — Kuros BioSciences B.V.
Locations (1):
- Orthopaedic Institute of Western Kentucky, Paducah, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No